CLINICAL TRIAL: NCT06503289
Title: Effects of The Removal of Myoglobin With CytoSorb on The Endothelium and Glycocalyx Shedding Biomarkers in Patients With Rhabdomyolysis
Brief Title: Myoglobin Removal With CytoSorb in Rhabdomyolysis
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Olcay Dilken, Anesthesiologist And Intensivist, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2346
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury; Rhabdomyolysis; Endothelial Dysfunction
Keywords: Myoglobin; Rhabdomyolysis; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury; Rhabdomyolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cytosorb therapy: 18 years older patients who need cytsorb therapy due to rhabdomyolysis
  Interventions: Device: Cytosorb therapy

INTERVENTIONS:
Device: Cytosorb therapy — Extracorporeal treatment with cytosorb filter to patients diagnosed with rhabdomyolysis

SUMMARY:
The aim of this observational study is to assess whether myoglobin removal with CytoSorb® ameliorates endothelial damage in severe rhabdomyolysis patients who are admitted to the intensive care unit. The primary objective of the study is:

- Does myoglobin removal with CytoSorb® reduces glycocalyx degradation markers?

Patients with severe rhabdomyolysis will receive the intervention and blood samples will be obtained in regular intervals.

DETAILED DESCRIPTION:
Rhabdomyolysis is characterized by destruction of muscle by various causes and is diagnosed by increased creatine kinase concentrations in the blood. Myoglobin released into the blood may cause acute kidney injury in up to half of these patients. The mortality caused by severe rhabdomyolysis is also high (32%). Extracorporeal modalities, such as CytoSorb (CS) can effectively eliminate the myoglobin from the bloodstream.

In addition to ischemic and inflammatory damage, myoglobin also causes direct endothelial cell injury. Degradation of the endothelial glycocalyx layer can be assessed by several biomarkers such as Syndecan-1, Heparan sulfate, cadherin

However, it is not fully known whether myoglobin elimination improves the outcomes or it is irrelevant of the outcome.

The investigator hypothesized that myoglobin elimination with CS alleviates the damage inflicted upon the endothelium and may have a role in improving patient outcomes in severe rhabdomyolysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Creatine Kinase > 5000 IU/L.
* Myoglobin results can be obtained only after 5 working days after sampling in our center, therefore it cannot be used as an inclusion criteria.
* GFR below 40 ml/min.

Exclusion Criteria:

* High dose vasopressor requirement
* Not expected to survive > 24 h
* Lack of consent to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years and older patients who need cytosorb therapy due to rhadomyolysis
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Syndecan-1 | 12 hour
  Reduction in Syndecan-1 with CS therapy

SECONDARY OUTCOMES:
glycocalyx markers | 12 hour
  Sustained reduction in other glycocalyx markers after CS therapy
myoglobin | 12 hours
  Reduction in myoglobin levels with CS therapy

CONTACTS AND LOCATIONS:
Overall Officials: mustafa altınay, Study Director — şişli etfal eğitim araştırma hastanesi
Locations (1):
- Sisli etfal research and training hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albrecht F, Schunk S, Fuchs M, Volk T, Geisel J, Fliser D, Meiser A. Rapid and Effective Elimination of Myoglobin with CytoSorb(R) Hemoadsorber in Patients with Severe Rhabdomyolysis. Blood Purif. 2024;53(2):88-95. doi: 10.1159/000534479. Epub 2023 Nov 2. PMID 37918366
- [Background] D'Agnillo F, Alayash AI. A role for the myoglobin redox cycle in the induction of endothelial cell apoptosis. Free Radic Biol Med. 2002 Oct 15;33(8):1153-64. doi: 10.1016/s0891-5849(02)01007-9. PMID 12374627
- [Background] Hahn RG, Patel V, Dull RO. Human glycocalyx shedding: Systematic review and critical appraisal. Acta Anaesthesiol Scand. 2021 May;65(5):590-606. doi: 10.1111/aas.13797. Epub 2021 Mar 7. PMID 33595101